CLINICAL TRIAL: NCT03200886
Title: Comparison of the Efficacy of Intra-articular Hybrid Hyaluronic Acid and Steroid in Patients With Rizoarthrosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, fioravanti antonella, Antonella Fioravanti, MD, PhD, Azienda Ospedaliera Universitaria Senese
Other Study IDs: COMB-IAL-V-TRIAM 01
Record Dates: First submitted 2017-06-14; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis Thumb
Keywords: hyaluronic acid; intra-articular injections; triamcinolone; osteoarthritis of the thumb
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sinovial H-L Group: The patients treated have received one cycle of two injections (at baseline and 15 days apart) of 1 ml of Sinovial H-L® (3.2% - 16mg + 16mg, Ibsa).
  Interventions: Device: Sinovial H-L
- Control Group: The patients have received two i.a. injections (at baseline and 15 days apart) of 0.5 ml of triamcinolone acetonide (Kenacort® 20 mg, Bristol-Myers Squibb Srl).
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Device: Sinovial H-L — Patients were treated with an hybrid form of hyaluronic acid (Sinovial H-L) obtained through thermo-chemical processes from the combination of high (1100-1400 kDa) and low (80-100 kDa) MW fractions.
  Groups: Sinovial H-L Group
Drug: Triamcinolone Acetonide — The patients have received two i.a. injections (at baseline and 15 days apart) of 0.5 ml of triamcinolone acetonide (Kenacort® 20 mg, Bristol-Myers Squibb Srl)
  Groups: Control Group

SUMMARY:
Osteoarthritis of the trapeziometacarpal joint (TMJ), also called rhizarthrosis is a common disease, mostly affecting post-menopausal women. Intra-articular therapy with hyaluronic acid (HA) was usually recommended as a second-line treatment after failure of non-pharmacological modalities, only in early stages of the disease .Aim of the present observational, retrospective, comparative study is the assessment of the efficacy and tolerability of i.a. injections of an hybrid HA formulation (Synovial H-L®) in comparison to triamcinolone in patients with TMJ Osteoarthritis (OA). We are analyzing the records collected in the departmental archives of outpatients affected by TMJ OA, according to the ACR criteria for the classification for hand OA and who were treated with i.a. Sinovial H-L or triamcinolone acetonide from December 1st, 2015 to December 1st 2016.The patient's assessment of spontaneous hand pain on a 0-100 mm VAS with 0 representing the absence of pain and the FIHOA score validated in Italian language were routinely recorded and documented in our centre prior to the injections (T0), at the time of the second i.a. administration (T1), after one month (T2) and after 3 (T3) and 6 months (T4) following the i.a. therapy.

The primary outcome criteria of our study is the change of VAS and FIHOA from baseline to the end of treatment. Furthermore, we chose as secondary outcomes the duration of morning stiffness, the Italian version of Health Assessment Questionnaire (HAQ) and the validated Italian version of the Medical Outcomes Study 36-Item Short Form (SF-36) routinary registered in our medical record before the i.a. therapy, at the end of the treatment and after 1, 3 and 6 months.

The chi square test, t test or Kruskal-Wallis test, as appropriated, will be used to evaluate differences between groups before i.a. treatment the clinical and demographical data.

Mixed-effects linear regression models will be used to evaluate temporal trends and differences in the two groups for specific outcomes: VAS pain, VAS stiffness, FIHOA and PCS and MCS from SF-36 questionnaires. In these types of statistical models, the effects of the covariates and their standard errors are correctly estimated taking into account the hierarchical structure of the data (i.e., patients and visits). For the compute of SF-36s Z score will be used mean and SD of U.S. general population. Data analysis will be performed using Stata vers 13.0 software. Descriptive statistics will be used to summarize data as frequencies (categorical variables) or mean +/-SD (continuous variables) as appropriate. P values <0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* clinical symptoms in the treated thumb for at least 3 months prior to the beginning of i.a. treatment with at least 30 mm on a 0-100 Visual Analogue Scale (VAS) and a Functional Index for Hand OA (FIHOA) score of at least 6
* radiographic evidence of TMJ OA within the previous 6 months with a radiological score of II-III (using the Kellgren method)

Exclusion Criteria:

* any inflammatory joint disease
* septic arthritis
* major trauma
* prior surgery of the hand, wrist, and elbow
* coagulation disorders
* severe comorbidity
* past therapy with chondroitin sulfate, glucosamine, diacerein, steroids by any route of administration
* i.a. injection of any joint with corticosteroids or HA during the previous 6 months

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients of both sex affected by TMJ OA
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of VAS | basal time; 2 weeks; 1 month; 3 months; 6 months
  0-100 mm VAS with 0 representing the absence of pain.
Change of FIHOA | basal time; 2 weeks; 1 month; 3 months; 6 months
  FIHOA validated in Italian language

SECONDARY OUTCOMES:
Change of duration of morning stiffness | basal time; 2 weeks;1 month; 3 months; 6 months
  measured in minutes
Change of Health Assessment Questionnaire (HAQ) | basal time; 2 weeks; 1 month; 3 months; 6 months
  Italian version of HAQ
Change of the Medical Outcomes Study 36-Item Short Form (SF-36) | basal time; 2 weeks; 1 month; 3 months; 6 months
  validated Italian version of SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tenti, MD, Principal Investigator — University of Siena
Locations (1):
- Azienda Ospedaliera Senese, Siena, Italy

REFERENCES:
- [Result] Zhang W, Doherty M, Leeb BF, Alekseeva L, Arden NK, Bijlsma JW, Dincer F, Dziedzic K, Hauselmann HJ, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Maheu E, Martin-Mola E, Pavelka K, Punzi L, Reiter S, Sautner J, Smolen J, Verbruggen G, Zimmermann-Gorska I. EULAR evidence based recommendations for the management of hand osteoarthritis: report of a Task Force of the EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). Ann Rheum Dis. 2007 Mar;66(3):377-88. doi: 10.1136/ard.2006.062091. Epub 2006 Oct 17. PMID 17046965
- [Result] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Result] Henrotin Y, Raman R, Richette P, Bard H, Jerosch J, Conrozier T, Chevalier X, Migliore A. Consensus statement on viscosupplementation with hyaluronic acid for the management of osteoarthritis. Semin Arthritis Rheum. 2015 Oct;45(2):140-9. doi: 10.1016/j.semarthrit.2015.04.011. Epub 2015 Apr 30. PMID 26094903
- [Result] Fioravanti A, Cantarini L, Chellini F, Manca D, Paccagnini E, Marcolongo R, Collodel G. Effect of hyaluronic acid (MW 500-730 kDa) on proteoglycan and nitric oxide production in human osteoarthritic chondrocyte cultures exposed to hydrostatic pressure. Osteoarthritis Cartilage. 2005 Aug;13(8):688-96. doi: 10.1016/j.joca.2005.03.006. PMID 15923130
- [Derived] Tenti S, Pascarelli NA, Giannotti S, Galeazzi M, Giordano N, Fioravanti A. Can hybrid hyaluronic acid represent a valid approach to treat rizoarthrosis? A retrospective comparative study. BMC Musculoskelet Disord. 2017 Nov 13;18(1):444. doi: 10.1186/s12891-017-1809-5. PMID 29132341